CLINICAL TRIAL: NCT04702542
Title: To Develop Methods for the Rehabilitation of Chronic Gastroduodenal Pathology (CGDP) in Schoolchildren in the Primary Health Care System.
Brief Title: To Develop Methods for the Rehabilitation of Chronic Gastroduodenal Pathology in Children.
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tashkent State Medical University (Tashkent Pediatric Medical Institute), Uzbekistan (Other)
Responsible Party: Principal Investigator, Turdieva Shokhida Tolkunovna, MD, МD, associate professor of the Department "Outpatient care", Tashkent State Medical University (Tashkent Pediatric Medical Institute), Uzbekistan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: TashkentPediatricMI-2
Record Dates: First submitted 2021-01-03; First posted 2021-01-11 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Gastritis Chronic; Gastroduodenitis; Peptic Ulcer; Duodenal Ulcer
Keywords: children; duodenal ulcer; gastritis; gastroduodenitis; Helicobacter pylori; oxygen therapy; rehabilitation; peptic ulcer; teenagers
MeSH Terms: conditions — Peptic Ulcer; Duodenal Ulcer; Gastritis

STUDY DESIGN:
Intervention Model Description: Comparison of 2 mutually comparable patient groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Enteral oxygen therapy for the improvement of children with chronic gastroduodenal pathology. (Experimental): Enteral oxygen therapy is prescribed for children with chronic gastroduodenal pathology during the recovery period, after inpatient treatment, for 14 days, every day, in the form of an oxygen cocktail. An oxygen cocktail is prepared on the basis of a pharmaceutical product using herbal ingredients. The patient takes a 200 ml oxygen cocktail. using a small spoon, during the daytime.
  Interventions: Drug: Enteral oxygen therapy

INTERVENTIONS:
Drug: Enteral oxygen therapy — Enteral oxygen therapy during the rehabilitation period of patients with CGDP.
  Other Names: Standard recreational activities for children after inpatient treatment.

SUMMARY:
The object of the study will be children and adolescents from 6 to 15 years old, living in the city of Tashkent and in the Tashkent region. We will study patients with various clinical forms of chronic gastroduodenal pathology (CGDP). The effect of enteral oxygen therapy in the recovery of patients with CGDP due to the positive effect of the active form of oxygen on the hematological system and on the regenerative processes in the gastrointestinal tract will be studied. At the same time, the effect of enteral oxygen therapy on enhancing the effectiveness of eradication therapy during the treatment of carrier Helicobacter pylori due to the neutralization of the products of urea hydrolysis around bacteria under the action of reactive oxygen species will be studied.

DETAILED DESCRIPTION:
In recent years, among the non-infectious diseases of children and adolescents, there has been an increase in many nosological forms of pathology of the gastrointestinal tract. Scientific works of recent years show that all over the world much attention is paid to the problem of timely prevention and improvement of chronic diseases of the gastroduodenal zone in children. This is mainly due to the fact that the incidence of diseases of the digestive system among schoolchildren is steadily increasing. In the clinical practice of gastroenterologists, it is often necessary to influence the regeneration processes in the gastroduodenal zone. The object of the study will be children and adolescents from 6 to 15 years old, living in the city of Tashkent and in the Tashkent region. We will study patients with various clinical forms of chronic gastroduodenal pathology (CGDP). The effect of enteral oxygen therapy in the recovery of patients with CGDP due to the positive effect of the active form of oxygen on the hematological system and on the regenerative processes in the gastrointestinal tract will be studied. At the same time, the effect of enteral oxygen therapy on enhancing the effectiveness of eradication therapy during the treatment of carrier Helicobacter pylori due to the neutralization of the products of urea hydrolysis around bacteria under the action of reactive oxygen species will be studied.

ELIGIBILITY:
Inclusion Criteria:

* children and adolescents aged 6 to 15 years;
* children with chronic gastroduodenal pathology: chronic gastritis, chronic gastroduodenitis, chronic duodenitis, gastric and intestinal ulcers of both sexes;
* children who have the opportunity to visit the clinic.

Exclusion Criteria:

* children under 6 years old and adolescents over 15 years old;
* children with chronic diseases of internal organs, except for the gastrointestinal tract;
* children with psychosomatic and neurological disorders;
* children in hospital;
* children with endocrine diseases;
* children who are allergic to eggs;
* children with blood diseases;
* children with cancer.

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 320 (Estimated)
Dates: Start 2022-04-30 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Initial clinical examination of children and adolescents at risk of CGDP. | 2 weeks
  A clinical examination of patients will be carried out, consisting of:
  identification of complaints - epigastric pain, dyspeptic symptoms - vomiting, panos, constipation, loss of appetite (oral questioning based on standard questions and scale HBSC (Health Behaviour in School-aged Children, A.King, 1996); collection of data on the presence in the family of a patient with this disease (oral survey based on standard questions); general examination of the patient - the presence of abdominal pain syndrome, stiffness of the abdominal muscles, intestinal distention (palpation, percussion, auscultation).
Identification of Helicobacter pylori infection. | 2 weeks
  The study for Helicobacter pylori (HP) infection will be based on the qualitative determination of the pathogen by two mutually unrelated methods: using a breath test (HELIK® test system with an indicator tube) and an immunochromatographic fecal sample for the presence of occult blood (erythrocyte cells).The interpretation of the test is either "positive" or "negative". The patient will be considered HP infected if both tests are positive.
Esofibrogastroduodenoscopy at the start of the study | 2 weeks
  Esofibrogastroduodenoscopy is carried out with an assessment of the endoscopic picture of the visible mucous membranes of the stomach and duodenum according to the criteria of the generally accepted Sydney classification (1990, with a modification of 1996), with a description of the visible mucous organ: the presence of areas of hyperemia, ulcers, atrophy, hypertrophy, scarring (visual description).
Treatment of identified patients. | 6 weeks
  If a disease is detected, the patient will be referred for treatment to a specialized children's hospital (Tashkent), where he will receive appropriate treatment according to generally accepted standards. The effectiveness of treatment will be assessed by the manifestation of clinical symptoms:
  the presence of complaints - epigastric pain, dyspeptic symptoms - vomiting, panos, constipation, loss of appetite (oral questioning based on standard questions); general examination of the patient - the presence of abdominal pain syndrome, stiffness of the abdominal muscles, intestinal distention (palpation, percussion, auscultation).
Rehabilitation of patients using enteral oxygen therapy. | 6 weeks
  Rehabilitation of children and adolescents with chronic gastroduodenal pathology after inpatient or outpatient treatment using enteral oxygen therapy is carried out. Studies will be conducted on the content in the peripheral blood in patients:
  hemoglobin (HGB, Hb, g/dL), erythrocytes (RBC, n x 1012/L), the content of hemoglobin in the erythrocyte (MCH, pg/cell), concentration in the erythrocyte of hemoglobin ( MCHC, g/dL).
  EFGDS is performed with an assessment of the endoscopic picture of the visible mucous membranes of the stomach and duodenum, according to the criteria of the generally accepted Sydney classification (1990, with a modification of 1996), with a description of the visible mucous organ: the presence of areas of hyperemia, ulcers, atrophy, hypertrophy, scarring.
Esofibrogastroduodenoscopy after rehabilitation. | 2 weeks
  After rehabilitation measures using enteral oxygen therapy, repeated esofibrogastroduodenoscopy (EFGDS) will be performed. EFGDS is carried out with an assessment of the endoscopic picture of the visible mucous membranes of the stomach and duodenum according to the criteria of the generally accepted Sydney classification (1990, with a modification of 1996), with a description of the visible mucous organ: the presence of areas of hyperemia, ulcers, atrophy, hypertrophy, scarring (visual description).

SECONDARY OUTCOMES:
Statistical data processing. | 8 weeks
  Statistical data processing will be carried out using Microsoft Excel 7.0 for Windows-XP, with the definition of the arithmetic mean (M) and standard deviation (s). When characterizing the statistical significance of the differences, the Student's t-test was used, with the determination of the limit of the confidence interval based on the Student's distribution table. The results will be assessed as statistically significant at a probability level of P <0.05. Comparison is made between groups of patients receiving enteral oxygen therapy and those not receiving.

CONTACTS AND LOCATIONS:
Overall Officials: Shokhida Turdieva, MD, Study Director — Tashkent State Medical University (Tashkent Pediatric Medical Institute), Uzbekistan
Locations (1):
- Tashkent Pediatric Medical Institute, Tashkent, Uzbekistan

IPD SHARING:
Plan to Share IPD: No
Joint study of the regenerative properties of oxygen in chronic pathology of the gastrointestinal tract.